CLINICAL TRIAL: NCT06155227
Title: Effect of Aerobic Exercise Combined With Blood Flow Restriction on Cardiopulmonary Function and Functional Activities in Frail Older Adults
Brief Title: Blood Flow Restriction With Aerobic Exercise in Frail Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Pei-Yun Lee, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-112-370
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Rehabilitation
Keywords: Blood flow restriction; Aerobic exercise; Frailty; Elderly
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: aerobic exercise combined with blood flow restriction
- Control Group (Active Comparator)
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise combined with blood flow restriction — aerobic exercise combined with blood flow restriction for 18 sessions
  Arms: Experimental Group
Other: aerobic exercise — aerobic exercise for 18 sessions
  Arms: Control Group

SUMMARY:
Background:Frailty is most often defined as a syndrome of physiological decline in late life, characterized by marked vulnerability to adverse health outcomes. Exercise intervention including aerobic exercise training has been proven to be effective in improving aerobic capacity and frail condition in elderly. Recently a novel training method using blood flow restriction (BFR) combined with aerobic exercise has shown positive effects on muscles strength and physical function in healthy elderly. This training method only required lower exercise intensity compared with traditional aerobic exercise to observe improvement. However, it is still unclear whether aerobic exercise training combined with BFR could also improve aerobic capacity and physical function in frail older adults. Therefore, the aim of this study will be to investigate the effect of aerobic exercise combined with BFR on cardiopulmonary function and functional activities in frail older adults.

Method: This study will be an assessor-blind randomized controlled trial.Participants aged over 65 years old with more than one item positive of Fried frailty phenotype assessment results will be recruited from the hospital and nearby communities. The participants will be randomly assigned to one of two training groups, aerobic exercise with BFR and only aerobic exercise. The exercise will be executed 30 minutes/session, three sessions/week for six weeks. Cardiopulmonary function and performance of functional activities will be assessed at pre-training, 3 weeks after training, post-training, and 3- and 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* more than one positive item of Fried frailty phenotype assessment
* able to walk more than 8 meters independently
* can understand and follow more than three-step order

Exclusion Criteria:

* severe hypertension (>160/100 mmHg)
* cardiovascular disease, such as myocardial infarction, New York Heart Association class III or IV heart failure, pulmonary hypertension
* deep vein thrombosis or peripheral vascular disease
* peripheral neuropathy due to diabetes
* neuromuscular diseases, such as stroke, Parkinson's disease, etc.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lower extremity muscle strength | Before training
  Use an hand-held dynamometer to measure bilateral lower limb muscle strength
Lower extremity muscle strength | After completing three-week training
  Use an hand-held dynamometer to measure bilateral lower limb muscle strength
Lower extremity muscle strength | After completing six-week training
  Use an hand-held dynamometer to measure bilateral lower limb muscle strength
Lower extremity muscle strength | At three weeks after completing the training
  Use an hand-held dynamometer to measure bilateral lower limb muscle strength
Lower extremity muscle strength | At six weeks after completing the training
  Use an hand-held dynamometer to measure bilateral lower limb muscle strength
Pulmonary function | Before training
  Pulmonary function includes tidal volume, vital capacity, forced vital capacity, and forced expiratory volume in one second
Pulmonary function | After completing three-week training
  Pulmonary function includes tidal volume, vital capacity, forced vital capacity, and forced expiratory volume in one second
Pulmonary function | After completing six-week training
  Pulmonary function includes tidal volume, vital capacity, forced vital capacity, and forced expiratory volume in one second
Pulmonary function | At three weeks after completing the training
  Pulmonary function includes tidal volume, vital capacity, forced vital capacity, and forced expiratory volume in one second
Pulmonary function | At six weeks after completing the training
  Pulmonary function includes tidal volume, vital capacity, forced vital capacity, and forced expiratory volume in one second
Timed up and go test | Before training
  This test measure the time taken by an individual to stand up from a chair , walk 3 meters, turn, walk back to the chair, and sit down
Timed up and go test | After completing three-week training
  This test measures the time taken by an individual to stand up from a chair , walk 3 meters, turn, walk back to the chair, and sit down
Timed up and go test | After completing six-week training
  This test measures the time taken by an individual to stand up from a chair , walk 3 meters, turn, walk back to the chair, and sit down
Timed up and go test | At three weeks after completing the training
  This test measure the time taken by an individual to stand up from a chair , walk 3 meters, turn, walk back to the chair, and sit down
Timed up and go test | At six weeks after completing the training
  This test measure the time taken by an individual to stand up from a chair , walk 3 meters, turn, walk back to the chair, and sit down
2 minutes step test | Before training
  Number of steps completed in 2 min
2 minutes step test | After completing three-week training
  Number of steps completed in 2 min
2 minutes step test | After completing six-week training
  Number of steps completed in 2 min
2 minutes step test | At three weeks after completing the training
  Number of steps completed in 2 min
2 minutes step test | At six weeks after completing the training
  Number of steps completed in 2 min
6 minutes walking test | Before training
  Record the distance walked in 6 minutes
6 minutes walking test | After completing three-week training
  Record the distance walked in 6 minutes
6 minutes walking test | After completing six-week training
  Record the distance walked in 6 minutes
6 minutes walking test | At three weeks after completing the training
  Record the distance walked in 6 minutes
6 minutes walking test | At six weeks after completing the training
  Record the distance walked in 6 minutes
Walking speed | Before training
  Test the gait speed under preferred and maximum speed walking
Walking speed | After completing three-week training
  Test the gait speed under preferred and maximum speed walking
Walking speed | After completing six-week training
  Test the gait speed under preferred and maximum speed walking
Walking speed | At three weeks after completing the training
  Test the gait speed under preferred and maximum speed walking
Walking speed | At six weeks after completing the training
  Test the gait speed under preferred and maximum speed walking

SECONDARY OUTCOMES:
Body composition | Before training
  Use Inbody 270 to measure skeletal muscle mass of the whole body and the four extremities
Body composition | After completing six-week training
  Use Inbody 270 to measure skeletal muscle mass of the whole body and the four extremities
Body composition | At three weeks after completing the training
  Use Inbody 270 to measure skeletal muscle mass of the whole body and the four extremities
Body composition | At six weeks after completing the training
  Use Inbody 270 to measure skeletal muscle mass of the whole body and the four extremities

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No